CLINICAL TRIAL: NCT02643381
Title: Etomidate Versus Ketamine for Emergency Endotracheal Intubation: a Prospective Randomized Clinical Trial
Acronym: EvK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Gerald Matchett, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022015-023
Record Dates: First submitted 2015-12-11; First posted 2015-12-31 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Cardiopulmonary Arrest; Respiratory Arrest
Keywords: etomidate; ketamine; endotracheal intubation; anesthesia induction medications
MeSH Terms: conditions — Heart Arrest; Apnea | interventions — Etomidate; Ketamine; Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etomidate (Experimental): Patients randomized to this group will receive etomidate immediately prior to emergency endotracheal intubation.
  Interventions: Drug: Etomidate; Procedure: Emergency Endotracheal Intubation; Device: Mechanical Ventilation
- Ketamine (Experimental): Patients randomized to this group will receive ketamine immediately prior to emergency endotracheal intubation.
  Interventions: Drug: Ketamine; Procedure: Emergency Endotracheal Intubation; Device: Mechanical Ventilation

INTERVENTIONS:
Drug: Etomidate — Patients randomized to this group will receive etomidate immediately prior to emergency endotracheal intubation.
  Arms: Etomidate
Drug: Ketamine — Patients randomized to this group will receive ketamine immediately prior to emergency endotracheal intubation.
  Arms: Ketamine
Procedure: Emergency Endotracheal Intubation — Patients enrolled in the study will be endotracheally intubated. (A breathing tube will be placed into the patient's mouth and trachea). This procedure is being done as part of standard emergency care. Standard endotracheal tubes will be used. Our hospital uses primarily Mallinckrodt (TM) brand endotracheal tubes.
Device: Mechanical Ventilation — Patients enrolled in the study will be mechanically ventilated, using a standard ventilator used in our hospital. The mechanical ventilator is attached to the patient's endotracheal tube and helps sustain the patient's life. Our hospital uses several brands of mechanical ventilators.

SUMMARY:
Patients who are having problems breathing sometimes require placement of a breathing tube in their mouth and windpipe. The purpose of this breathing tube is to save the patient's life. It is common to give the patient a medication to sedate him or her before the breathing tube is placed. For patients who are gravely ill two medications are commonly used: etomidate or ketamine. Both medications have risks and benefits. Researchers at UT-Southwestern Medical Center and Parkland Memorial Hospital would like to do a study to figure out which one is better for our patients.

DETAILED DESCRIPTION:
Critically ill individuals who require emergency endotracheal intubation (placement of a breathing tube in the patient's mouth) usually require sedation or anesthesia to make this process tolerable. There are several medication choices for anesthesia, including medications like etomidate, ketamine and propofol. Of these, etomidate and ketamine are frequently used for critically ill patients because they have minimal effects on the patient's vital signs (blood pressure and heart rate). Both etomidate and ketamine are standard-of-care medications, locally and nationally, and both are frequently used to sedate a patient for this procedure. Both etomidate and ketamine have potential side effects. One of the potential side effects of etomidate is suppression of adrenal gland function. It is not known if this affects patients' outcomes in significant ways. One of the potential side effects of ketamine is a slight increase in patients' heart rates. It is not known if this affects patients' outcomes in significant ways.

The EvK Trial will be conducted at Parkland Memorial Hospital by investigators in the Departments of Anesthesiology, Emergency Medicine, Medicine / Critical Care Medicine, Surgery, and Pharmacy. The study will randomize critically ill patients who require emergency endotracheal intubation to one of two groups: Etomidate or Ketamine. We will observe the patients' outcomes. The only study intervention involves randomizing individual patients to one medication or the other. All study follow-up beyond that point is done by review of medical records.

Because of the nature of this study - an emergency procedure on a critically ill patient - the study will require institutional review board permission not to obtain written informed consent from the patient prior to randomization of study drug for administration for endotracheal tube placement. Prior to enrollment of patients the study team will carry out a comprehensive Community Consultation Plan, which is designed to inform the community about the research study. This is in accordance with rules set forth by the U.S. Food and Drug Administration (FDA 21 CFR 50.24).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (male or female) requiring emergency endotracheal intubation.

Exclusion Criteria:

* Children (<18 years old).
* Women who are known to be pregnant.
* Any patient who has been previously randomized in the EvK Trial.
* Patients who require endotracheal intubation without sedative medication. For example, patients in full cardiac arrest.
* Patients with a known allergy to ketamine or etomidate.
* Any individual wearing a MedAlert bracelet indicating that he/she has formally opted out of the EvK Trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Matchett, MD, Principal Investigator — University of Texas
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate anonymous data will be published in accord with our IRB approval.

REFERENCES:
- [Result] Matchett G, Ryan TJ, Sunna MC, Lee SC, Pepe PE; EvK Clinical Trial Group. Measuring the cost and effect of current community consultation and public disclosure techniques in emergency care research. Resuscitation. 2018 Jul;128:37-42. doi: 10.1016/j.resuscitation.2018.04.033. Epub 2018 Apr 30. PMID 29715485
- [Derived] Matchett G, Gasanova I, Riccio CA, Nasir D, Sunna MC, Bravenec BJ, Azizad O, Farrell B, Minhajuddin A, Stewart JW, Liang LW, Moon TS, Fox PE, Ebeling CG, Smith MN, Trousdale D, Ogunnaike BO; EvK Clinical Trial Collaborators. Etomidate versus ketamine for emergency endotracheal intubation: a randomized clinical trial. Intensive Care Med. 2022 Jan;48(1):78-91. doi: 10.1007/s00134-021-06577-x. Epub 2021 Dec 14. PMID 34904190

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etomidate | Ketamine
Started | 400 | 401
Completed | 396 | 395
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etomidate | Ketamine | Total
Number analyzed (Participants) | 396 | 395 | 791
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (15.2) | 55.4 (16.0) | 55.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 150 | 303
  Male | 243 | 245 | 488
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 250 | 246 | 496
  Black | 133 | 122 | 255
  Other | 13 | 27 | 40
  Hispanic | 141 | 139 | 280
Region of Enrollment [Number; unit: participants]
  United States | 396 | 395 | 791

OUTCOME MEASURES:

1. Primary Outcome: Survival at Day 7
Description: Survival is defined as the number of participants survived at day 7 following emergency endotracheal intubation
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
Participants | 306 | 336

2. Secondary Outcome: Survival at Day 28
Description: Survival is defined as the number of participants survived at day 28 following emergency endotracheal intubation
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
Participants | 254 | 264

3. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Scores
Description: Sequential Organ Failure Assessment (SOFA) is a scoring system that assesses the performance of several organ systems. Possible scores range from 0 to 24. Higher score indicates higher degree of organ dysfunction
Time Frame: Day 1, Day 2, Day 3, Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
score on a scale
  Day 1 | 10.7 (4.6) | 10.9 (4.5)
  Day 2 | 9.8 (5.1) | 9.5 (4.9)
  Day 3 | 8.4 (5.3) | 8.4 (5.1)
  Day 4 | 7.4 (5.2) | 7.4 (5.4)

4. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration (in days) from insertion to removal of mechanical ventilation
Time Frame: From time of documented insertion until the time of documented removal, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
Days | 5 [3 to 9] | 5 [3 to 10]

5. Secondary Outcome: Duration of Catecholamine Therapy
Description: Time (in days) from start to end of catecholamine therapy
Time Frame: From time of documented start of therapy until the time of documented end of therapy, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
Days | 1 [0 to 3] | 1 [0 to 3]

6. Secondary Outcome: Length of Stay in ICU
Description: Length (in days) of ICU stay
Time Frame: Assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
Days | 8 [4 to 16] | 9 [5 to 14]

7. Secondary Outcome: Number of Participants With New Diagnosis of Adrenal Insufficiency
Description: New diagnosis of adrenal insufficiency will be assessed by the the primary treating medical or surgical team via chart review
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 396 | 395
Participants | 11 | 4

8. Secondary Outcome: Number of Attempts Necessary to Intubate
Description: This referrers to the number of documented intubation attempts necessary to intubate the patient.
Time Frame: Immediate (Day 1)
Population: Clinical information incomplete or missing from 5 patients randomized to Etomidate and 6 patients randomized to Ketamine.
Measure: Count of Participants; unit: Participants
Arm/Group | Etomidate | Ketamine
Number analyzed (Participants) | 391 | 389
Participants
  1 Attempt (successfully intubated) | 357 | 355
  2 Attempts (successfully intubated) | 29 | 26
  3 or More Attempts (successfully intubated) | 4 | 5
  Surgical Airway | 1 | 3

ADVERSE EVENTS:
Time Frame: Day 1-28
Description: Adverse study-related events
Arm/Group | Etomidate | Ketamine
All-Cause Mortality (participants affected / at risk) | 142/396 | 131/395
Serious Adverse Events (participants affected / at risk) | 10/396 | 9/395
Other Adverse Events (participants affected / at risk) | 0/396 | 0/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etomidate (N=396) | Ketamine (N=395)
Oral/ dental trauma (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) — Trauma noted in narrative form in clinical documentation.
Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) — Bleeding noted in narrative form in clinical documentation.
Aspiration (Injury, poisoning and procedural complications) | 8 (8) | 2 (2) — Aspiration noted in narrative form in clinical documentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT02643381/Prot_SAP_001.pdf